CLINICAL TRIAL: NCT05321823
Title: Improving Access to Breast Cancer Screening and Treatment in Nigeria: The Triple Mobile Assessment and Patient Navigation Model
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Obafemi Awolowo University (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Adeleye Omisore, Dr., Obafemi Awolowo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: ERC/2020/10/11 (26/10/2020); #60303257 (Other Grant/Funding Number: Pfizer Inc.)
Record Dates: First submitted 2022-03-24; First posted 2022-04-11 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Breast Cancer
Keywords: Screening; Treatment; Navigation; Triple Mobile assessment
MeSH Terms: conditions — Breast Neoplasms | interventions — Ultrasonography, Mammary; Mammography

STUDY DESIGN:
Intervention Model Description: The study will be carried out in 2 local counties (Local Government Areas) in Osun State, South-West, Nigeria, Ife North Local County and Ife East Local County. Three districts in Ife North Local County with an estimated screening population (women 40-70 years) of 5,800 will be randomly selected to serve as the intervention community, while 2 districts in Ife East Local County with an estimated screening population of 4,500 will be randomly selected to serve as the control community. Both communities will receive awareness and education, but only the intervention community will receive screening and navigation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Control (No Intervention): Two districts in Ife East Local County with an estimated screening population of 4,500 will be randomly selected to serve as the control community. The control arm will not receive iBE screening and clinical breast examinations by the community health nurses and nor get navigated to have ultrasound, mammography, biopsy and referral for treatment to the tertiary hospital if indicated within their community. All women for screening and diagnostic workup in the control community will be directed to the tertiary hospital to receive breast care.
- Intervention (Experimental): Three districts in Ife North Local County with an estimated screening population (women 40-70 years) of 5,800 will be randomly selected to serve as the intervention community. Women in the intervention community will receive iBreast and clinical breast examinations by the community health nurses and get navigated to have ultrasound, mammography, biopsy and referral for treatment to the tertiary hospital if indicated within their community.
  Interventions: Device: iBreast device; Other: Clinical Breast Examination; Diagnostic Test: Breast ultrasound; Diagnostic Test: Mammography

INTERVENTIONS:
Device: iBreast device — The iBreast (iBE) device is an automated, battery powered, portable device designed to be used by community health nurses as a screening and triage tool. The iBE is designed to be used by a community health worker or lay person after appropriate training. In resource-limited settings, it potentially provides an easily accessible, low-cost method to assess the breast for findings that warrant further evaluation.
  Other Names: UE Life Sciences Inc.
  Arms: Intervention
Other: Clinical Breast Examination — The standard clinical breast examination (CBE) will be performed by the community health nurses in the selected primary health care centers where patients will present for screening or diagnostic workup in the intervention community
  Other Names: CBE
  Arms: Intervention
Diagnostic Test: Breast ultrasound — Women in the intervention community who have positive iBE and/or CBE findings will be navigated by the community health nurses to have ultrasound with or without ultrasound-guided breast biopsy if indicated by the radiologist using portable ultrasound tablets that will be brought to the intervention community.
  Arms: Intervention
Diagnostic Test: Mammography — Women in the intervention community who have positive iBE and/or CBE findings will be navigated by the community health nurses to have mammography done using a mobile mammography van that will be brought to the intervention community.
  Arms: Intervention

SUMMARY:
The goal of this study is to establish a novel community-based breast cancer program to address delayed presentation and lack of access to diagnostic and treatment facilities in South-West Nigeria. It is aimed at evaluating the impact of a novel breast cancer early detection program using triple mobile assessment (innovative handheld iBreast Exam [iBE] device, mobile ultrasound, and mobile mammography) and patient navigation program in a Nigerian community.

DETAILED DESCRIPTION:
This study aims to provide screening to asymptomatic women 40-70 years and to provide diagnostic evaluation to women 30-70 years presenting with breast symptoms in a community in South-West Nigeria.

The project will use a cluster randomized design with 1 community serving as the intervention arm and another community serving as the control arm. Both communities will receive breast cancer awareness and education but only the intervention community will receive screening, mobile imaging and navigation. Screening with targeted clinical history, Clinical Breast Exam (CBE), and iBE will be performed by trained Community Health Nurses in the intervention community. Women with positive CBE or iBE findings will undergo breast imaging with mobile mammography and portable ultrasound, as well as biopsy when indicated by the Radiologist who visits the community once a month, and receive navigation by the nurses to the point of care. The control population will receive breast cancer awareness without an organized screening, imaging or navigation program. Women presenting to the Primary Health Care Centers in the control community will be referred to the Teaching Hospital as per current standard of care. Record of all breast cancer cases seen in the 2 communities during the study period will be obtained.

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic women 40 - 70 years
* Symptomatic women (with breast-related symptoms) 30 - 70 years

Exclusion Criteria:

* Male subjects
* Women living outside the study locations (Ife East and Ife North districts)

Ages: 30 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — The study is addressing breast cancer screening and treatment in women
Enrollment: 4100 (Estimated)
Dates: Start 2021-12-08 (Actual); Primary Completion 2023-10-31 (Estimated); Study Completion 2023-10-31 (Estimated)

PRIMARY OUTCOMES:
Participation rate | After year 1 of the 2-year study period
  Percentage of women screened of the total number of eligible women in each community.
Abnormal call rate | After year 1 of the 2-year study period
  Number of women with abnormalities detected on iBE and/or CBE requiring further evaluation either by imaging or biopsy out of the total number of women screened.
Breast cancer detection rate | After year 1 of the 2-year study period
  Number of histologically diagnosed cases of breast cancer per 1,000 screened populations.
Stage at presentation | After year 1 of the 2-year study period
  The tumour, node and metastasis (TNM) stage among those with histologically confirmed breast cancer.
Timeline from presentation to treatment | After year 1 of the 2-year study period
  Time interval between presentation for screening in the community and treatment in the tertiary hospital
Retention rate | After year 2 of the 2-year study period
  Number of women who return for repeat annual screening of the total initial number of women screened.

CONTACTS AND LOCATIONS:
Overall Officials: Adeleye D Omisore, MBBS, M.Sc, FWACS, FMCR, Principal Investigator — Obafemi Awolowo University
Locations (1):
- Obafemi Awolowo University Teaching Hospitals Complex, Ile-Ife, Osun State, Nigeria

IPD SHARING:
Plan to Share IPD: Yes
The study protocol, statistical analysis plan, and informed consent form will be made available on clinicaltrials.gov if and when required. With study data being uploaded to redcap hosted by the sponsor organization (Obafemi Awolowo University), de-identified individual participant data can be made available under the terms of a data use agreement 12 moths after publication of study results.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data can be available beginning 12 months after publication of the study results up to to 36 months post publication.
Access Criteria: Researchers with approved proposals

REFERENCES:
- [Derived] Omisore AD, Olasehinde O, Wuraola FO, Sutton EJ, Sevilimedu V, Omoyiola OZ, Romanoff A, Owoade IA, Olaitan AF, Kingham TP, Alatise OI, Mango VL. Improving access to breast cancer screening and treatment in Nigeria: The triple mobile assessment and patient navigation model (NCT05321823): A study protocol. PLoS One. 2023 Jun 13;18(6):e0284341. doi: 10.1371/journal.pone.0284341. eCollection 2023. PMID 37310983